CLINICAL TRIAL: NCT05994872
Title: A Randomized Controlled Trial of Reverse Drilling Technique in Improving Outcomes After Arthroscopic Anterior Cruciate Ligament Reconstruction: a Prospective, Multicenter, Single-blind, Randomized Controlled Surgical Trial
Brief Title: Reverse Drilling Technique in Improving Outcomes After Arthroscopic Anterior Cruciate Ligament Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo Medical Center Lihuili Hospital (Other Government); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Shaoxing Traditional Chinese Medicine Hospital (Unknown); Lishui Municipal Central Hospital (Other Government); The First People's Hospital of Huzhou (Other); Jiande First People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-0562
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Reverse drilling technique; Anterior cruciate ligament reconstruction; Tendon-to-bone healing
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Surgical doctor team, patient, outcome assessor, data analyst and image reviewer are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional extraction drilling (Sham Comparator): A standard hamstring autograft procedure was performed using traditional extraction drilling to prepare bone tunnel (n = 108).
  Interventions: Procedure: Traditional extraction drilling
- Reverse drilling technique (Experimental): A standard hamstring autograft procedure was performed using reverse drilling technique to prepare bone tunnel (n = 108).
  Interventions: Procedure: Reverse drilling technique

INTERVENTIONS:
Procedure: Reverse drilling technique — A standard hamstring autograft procedure was performed using reverse drilling technique to prepare bone tunnel.
  Arms: Reverse drilling technique
Procedure: Traditional extraction drilling — A standard hamstring autograft procedure was performed using traditional extraction drilling to prepare bone tunnel.
  Arms: Traditional extraction drilling

SUMMARY:
Anterior cruciate ligament (ACL) injuries and bone tunnel enlargement (BTE) after ACL reconstruction (ACLR) remain frequent issues. Bone dust (BD) produced by tunnel preparation with osteogenic ability and reverse drilling (RD), an easy compaction technique, make it accessible to enhance tendon-bone healing in ACLR. We hyposize that RD and BD synergistically improve outcomes after arthroscopic ACLR by improving peritunnel bone and preventing BTE.

DETAILED DESCRIPTION:
Compaction technique can create a denser bone tunnel wall with more cancellous bone autografting in situ by sequentially compressing cancellous bone trabeculae to bone tunnel walls, in contrast to conventional extraction reaming by which an enlarged gap is created and initial direct integration is limited between implants and bone, as chunks of cancellous bone are torn out, thereby being removed outside the tunnel. Biologically, a compaction technique was reported to increase the bone volume around grafts and provide a larger area of bone-to-graft contact for bone integration because of the spring-back effect. Mechanically, compaction of the bone graft into the femoral tunnel was reported to significantly increase stiffness of the grafts. Reverse drilling (RD) can compress peritunnel bone at the time of bone tunnel preparation to make the tunnel wall denser and smoother in comparison with extraction drilling (ED), reverse drilling yields the same compaction effect as the compaction technique. Bone dust (BD) is commonly defined as pieces of bone produced by a power-driven tool. It is universally accepted that bone debris more than 200 mm in particle size is classified as particulate bone and that bone debris no more than 200 mm is classified as BD. When applied for ACLR, BD could fully utilize the advantages of an autologous bone graft while avoiding invasive and traumatic bone harvesting procedures, as bone tunnel preparation is accompanied by the production of a considerable amount of BD. Therefore, BD grafting is promising for improving tendon-bone healing with safety and simplification. We refer to the technique of retaining BD in the bone tunnel after RD as the reverse drilling technique. We hyposize that reverse drilling technique can improve outcomes after arthroscopic anterior cruciate ligament reconstruction by improving peritunnel bone and preventing bone tunnel enlargement.

ELIGIBILITY:
Inclusion Criteria:

Patients with definite anterior cruciate ligament injuries on imaging or intraoperative arthroscopy (Sherman grading II and III), plan surgery within 45 days from injury; have basic literacy skills and unimpeded communication; have a smartphone and are able to use WeChat; and have been given informed consent and have signed to obtain an informed consent form, and the process must be in accordance with GCP requirements.

Exclusion Criteria:

1) Combined with other knee injuries (posterior cruciate ligament injury, patellar dislocation, osteoarthritis, etc.); 2) Suffering from systemic immune diseases; 3) Presence of other diseases or inflammatory diseases of the knee, including osteoarthritis, cervical spondylosis, rheumatoid arthritis, fibromyalgia, and rheumatic polymyalgia, etc.; 4) Patients who have had localized hormone injection therapy within 3 months; 5) Those who have participated in a clinical trials or are undergoing other clinical trials; 6) Those with severe primary cardiovascular lesions, pulmonary diseases, endocrine and metabolic diseases or serious diseases affecting their survival, such as tumors or AIDS, which in the opinion of the investigator are not suitable for enrollment; 7) Those with severe hepatic lesions, renal lesions, and hematologic lesions, such as renal function exceeding the upper limit of normal values and hepatic function exceeding two times the upper limit of normal values; and 8) Those with viral hepatitis, infectious diseases, severe abnormalities of coagulation mechanism and other diseases that the investigator considers inappropriate for surgery; 9) Pregnant or lactating women, or those who plan to conceive during the follow-up period, with a positive result of urinary human chorionic gonadotropin test prior to sampling; menstruating women should wait until the end of their menstruation period to undergo the surgery; 10) Patients with severe neurological or psychiatric disorders; 11) Those with a suspected or confirmed alcoholic substance abuse history; 12) Vulnerable groups: mentally ill, critically ill patients, pregnant women, illiterate, minors, cognitively impaired.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
IKDC Subjective Score | Patients will be followed up regularly at 3, 6, 9, 12, and 24 months after surgery.
  This table consists of knee joint assessment (10 items) and knee ligament examination (8 items), which includes joint pain, exercise level, and daily activity ability, with a total score of 0-100 points.
Bone tunnel enlargement | Patients will be followed up regularly at 3, 6, 9, 12, and 24 months after surgery.
  Measurement of bone tunnel enlargement through postoperative image

SECONDARY OUTCOMES:
Instrumented AP Knee Laxity | Patients will be followed up regularly at 3, 6, 9, 12, and 24 months after surgery.
  Arthrometer testing (KT-1000; MEDMetric) was used to measure the anterior displacement of the tibia with respect to the femur under 130 N of applied anterior force and performed in duplicate on each leg.

CONTACTS AND LOCATIONS:
Overall Officials: Haobo Wu, MD, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (6):
- China (6):
  - The First People's Hospital of Huzhou, Huzhou, Zhejiang
  - Lishui Municipal Central Hospital, Lishui, Zhejiang
  - Jiande First People's Hospital, Meicheng, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Shaoxing Traditional Chinese Medicine Hospital, Shaoxing, Zhejiang
  - Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoogeslag RAG, Huis In 't Veld R, Brouwer RW, de Graaff F, Verdonschot N. Acute Anterior Cruciate Ligament Rupture: Repair or Reconstruction? Five-Year Results of a Randomized Controlled Clinical Trial. Am J Sports Med. 2022 Jun;50(7):1779-1787. doi: 10.1177/03635465221090527. Epub 2022 Apr 29. PMID 35486517
- [Result] Murray MM, Fleming BC, Badger GJ; BEAR Trial Team; Freiberger C, Henderson R, Barnett S, Kiapour A, Ecklund K, Proffen B, Sant N, Kramer DE, Micheli LJ, Yen YM. Bridge-Enhanced Anterior Cruciate Ligament Repair Is Not Inferior to Autograft Anterior Cruciate Ligament Reconstruction at 2 Years: Results of a Prospective Randomized Clinical Trial. Am J Sports Med. 2020 May;48(6):1305-1315. doi: 10.1177/0363546520913532. Epub 2020 Apr 16. PMID 32298131
- [Result] Beard DJ, Davies L, Cook JA, Stokes J, Leal J, Fletcher H, Abram S, Chegwin K, Greshon A, Jackson W, Bottomley N, Dodd M, Bourke H, Shirkey BA, Paez A, Lamb SE, Barker K, Phillips M, Brown M, Lythe V, Mirza B, Carr A, Monk P, Morgado Areia C, O'Leary S, Haddad F, Wilson C, Price A; ACL SNNAP Study Group. Rehabilitation versus surgical reconstruction for non-acute anterior cruciate ligament injury (ACL SNNAP): a pragmatic randomised controlled trial. Lancet. 2022 Aug 20;400(10352):605-615. doi: 10.1016/S0140-6736(22)01424-6. PMID 35988569
- [Result] Fauno P, Kaalund S. Tunnel widening after hamstring anterior cruciate ligament reconstruction is influenced by the type of graft fixation used: a prospective randomized study. Arthroscopy. 2005 Nov;21(11):1337-41. doi: 10.1016/j.arthro.2005.08.023. PMID 16325084
- [Result] Weber AE, Delos D, Oltean HN, Vadasdi K, Cavanaugh J, Potter HG, Rodeo SA. Tibial and Femoral Tunnel Changes After ACL Reconstruction: A Prospective 2-Year Longitudinal MRI Study. Am J Sports Med. 2015 May;43(5):1147-56. doi: 10.1177/0363546515570461. Epub 2015 Feb 13. PMID 25681503
- [Result] Yang W, Li C, Ji X, Yao M, Hong J, Qu Z, Liu A, Wu H. Synergistic Effect of Reverse Drilling and Bone Dust on Femoral Tendon-Bone Healing After Anterior Cruciate Ligament Reconstruction in a Rabbit Model. Am J Sports Med. 2022 Dec;50(14):3844-3855. doi: 10.1177/03635465221129267. Epub 2022 Nov 3. PMID 36326437